CLINICAL TRIAL: NCT01022255
Title: Phase I Study of an Autologous Recombinant Idiotypic Vaccine Manufactured by magnICON® Technology for the Treatment of Patients With Relapsed or Transformed Follicular Lymphoma
Brief Title: Autologous Vaccine for Follicular Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Icon Genetics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMP0025-01
Record Dates: First submitted 2009-11-30; First posted 2009-12-01 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Lymphoma, Follicular
Keywords: autologous vaccine; follicular lymphoma; magnICON; plant-made vaccines; immune response
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Biological: Autologous FL vaccine

INTERVENTIONS:
Biological: Autologous FL vaccine — 1.0 mg of vaccine subcutaneously (s.c.) on Day 1, and followed by 125 µg GM-CSF s.c. at Day 1 -4, monthly until 8th vaccination, bimonthly until 12th vaccination (month 16)

SUMMARY:
This phase I study will evaluate the safety and tolerability of an autologous idiotype vaccine manufactured by magnICON technology for patients with relapsed follicular lymphoma who are in complete or partial remission following non-antiCD20 containing salvage therapy. Data in terms of idiotype-specific immune responses will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically proven follicular lymphoma (grade 1, 2, or 3a), in clinical relapse/progression requiring treatment
* Subjects must have had first line treatment consisting of rituximab with or without rituximab maintenance therapy (i.e. rituximab monotherapy, R-CHOP, R-CVP, R-FND, etc)
* At least 4 months since last rituximab exposure
* Subjects may have had any number of prior treatment regimens. If enrolled with transformed follicular lymphoma, study subject must have had anthracycline in a previous regimen
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Life expectancy of at least 12 months
* Presence of at least a 2x2 cm in diameter lymph node (either a single lymph node or combined volume of lymphoid tissue) accessible for excision; for histological confirmation of diagnosis and for manufacture of the vaccine
* Measurable disease in neck, chest, abdomen, or pelvis as assessed by computed tomography (CT) scan such that response to 2nd line chemotherapy can be defined by the criteria of Cheson et al (JCO 2007; 25:579, see appendix 15.2 and ref 65). PET scan results are not required for enrollment

Exclusion Criteria:

* Exposure to rituximab or antiCD-20 directed therapy within the 4 months prior to enrollment
* History of human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection
* Active clinically serious infections (> grade 2 National Cancer Institute Common Toxic Criteria [NCI-CTC] version 3.0)
* Symptomatic metastatic brain or meningeal tumors including lymphoma unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry
* History of organ allograft
* Patients undergoing renal dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with toxicities as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI/CTCAE) version 3.0 grade >/= 3 to the magnICON generated idiotype (Id) vaccine | One month after sixth vaccination (=7 month after achievement of tumour remission and recovery of normal blood values)

SECONDARY OUTCOMES:
Assessment of humoral idiotype-specific immune responses | One month after sixth vaccination (=7 month after achievement of tumour remission and recovery of normal blood values)
Assessment of cellular idiotype-specific immune responses | One month after sixth vaccination (=7 month after achievement of tumour remission and recovery of normal blood values)
Long-term safety/tolerability as determined by the proportion of patients with toxicities as assessed by the FDA CBER Guidance for Industry Toxicity Grading Scale in Preventive Vaccine Clinical Trials and the NCI/CTCAE version 4.02 grade >/= 3 | Up to the conclusion of a 12 cycle vaccination phase (month 16)

CONTACTS AND LOCATIONS:
Overall Officials: Company Study Director, Study Director — Icon Genetics
Locations (2):
- United States (2):
  - Burbank, California
  - Dallas, Texas